CLINICAL TRIAL: NCT00339014
Title: A Dose Parallel, Randomized, Placebo-Controlled, Multicenter Study of the Safety and Efficacy of Multiple Regimens of the Combination of Zonisamide CR Plus Bupropion SR in the Treatment of Subjects With Uncomplicated Obesity
Brief Title: Safety and Efficacy of Different Combinations of Zonisamide-CR Plus Bupropion-SR to Treat Uncomplicated Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Ronald Landbloom, MD, Orexigen Therapeutics, Inc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZB 201
Record Dates: First submitted 2006-06-18; First posted 2006-06-20 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Group 1 (Active Comparator): Zonisamide SR 120 mg/day plus Bupropion SR 280 mg/day
  Interventions: Drug: Zonisamide CR and Bupropion SR
- Group 2 (Active Comparator): Zonisamide SR 120 mg/day plus Bupropion SR 360 mg/day
  Interventions: Drug: Zonisamide CR and Bupropion SR
- Group 3 (Active Comparator): Zonisamide SR 240 mg/day plus Bupropion SR 280 mg/day
  Interventions: Drug: Zonisamide CR and Bupropion SR
- Group 4 (Active Comparator): Zonisamide SR 240 mg/day plus Bupropion SR 360 mg/day
  Interventions: Drug: Zonisamide CR and Bupropion SR
- Group 5 (Active Comparator): Zonisamide SR 360 mg/day plus Bupropion SR 280 mg/day
  Interventions: Drug: Zonisamide CR and Bupropion SR
- Group 6 (Active Comparator): Zonisamide SR 360 mg/day plus Bupropion SR 360 mg/day
  Interventions: Drug: Zonisamide CR and Bupropion SR
- Group 7 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Zonisamide CR and Bupropion SR — Zonisamide SR and Bupropion SR
  Arms: Group 1; Group 2; Group 3; Group 4; Group 5; Group 6
Other: Placebo — Identical placebo
  Arms: Group 7

SUMMARY:
The purpose of this study is to determine which of seven combinations of Zonisamide CR and Bupropion SR gives the best weight loss and is safe and well tolerated for the treatment of obesity not associated with the complications of obesity such as diabetes. In a previous study, the combination of zonisamide and bupropion SR was shown to be effective for weight loss compared to either zonisamide, bupropion SR alone or placebo. It is thought that by adjusting the doses of each drug, giving zonisamide in a controlled release (CR) form and increasing the doses more slowly, more weight loss and less side effects can be attained.

DETAILED DESCRIPTION:
Over the past few years, knowledge of the pathways and neural circuits that sense body energy stores has increased dramatically. In particular, it has been shown that the melanocortin system, a group of neuronal circuits in the arcuate nucleus of the hypothalamus, is the "final common pathway" for most energy state signals, and that melanocortin signaling is necessary for normal control of food intake and energy expenditure. Stimulation of POMC neurons by serotonergic and dopaminergic agents results in release of α-, β- and γ-MSH through the action of prohormone convertase-2 with a consequent decrease in appetite.A second counter-regulatory system that inhibits POMC activation is β-endorphin, which binds to a mu-opioid receptor (MOP-R) and acts as an auto-inhibitory "brake" on the activity of the melanocortin circuits. Bupropion is an approved antidepressant that blocks reuptake of serotonin and dopamine. This stimulates secretion of both α -MSH and β-endorphin. α -MSH binds to melanocortin receptors which in turn results in appetite suppression and increased energy expenditure. β-endorphin, however, binds to a mu-opioid receptor (MOP-R) and inhibits the activity of the melanocortin circuits. Zonisamide has multiple effects that may protect against seizures, including blockade of sodium channels, and reducing voltage dependent inward (T type) calcium currents, leading to neuronal stabilization. In addition to these actions, however, it is known to increase 5-hydroxytryptophan and dopamine levels, simultaneously stimulating α -MSH release while inhibiting AGRP release. Thus, the combination of bupropion and zonisamide stimulates the melanocortin system while blocking an important feedback inhibitory pathway.

The combination of zonisamide 400 mg/day and bupropion SR 300 mg/day has been shown to be more effective for weight loss than either monotherapy or placebo in subjects with uncomplicated obesity. The hypothesis for the current trial is that greater efficacy and improved tolerability can be achieved by adjusting the doses and titration of both bupropion SR and zonisamide, and by giving zonisamide in a controlled release (CR) formulation.

ELIGIBILITY:
Inclusion Criteria:

* Have body mass index (BMI) of 30 to 43 kg/m2
* Free from any other clinically significant illness or disease as determined by medical history and physical examination
* Non-smoker and no use of tobacco or nicotine products for at least 6 months prior to screening
* Normotensive (systolic <140 mm Hg; diastolic <90 mm Hg). Anti-hypertensive medications are allowed with the exception of adrenergic blockers, beta-blockers and clonidine. Medical regimen must be stable for at least 6 weeks
* LDL cholesterol < 190 mg/dL and triglycerides < 400 mg/dL. Medications for treatment of dyslipidemia are allowed as long as medical regimen has been stable for at least 6 weeks
* Negative serum pregnancy test in women with an intact uterus
* Score < 15 for depression and score < 15 for anxiety on Hospital Anxiety and Depression Scale (HADS)
* No clinically significant abnormality on ECG
* Not on eExcluded concomitant medications
* If female with intact uterus, be non-lactating, and agree to use effective contraception throughout the study period and for 30 days after discontinuation of study drugs.
* Able to comply with all required study procedures and schedule
* Able to use and have access to a touch tone telephone and to speak and read English

Exclusion Criteria:

* Obesity of known endocrine or genetic origin
* Serious medical condition
* Serious psychiatric illness
* Active suicidal ideation; score > 2 on the Mood Assessment questionnaire
* A response to Bipolar Disorder questions indicating the presence of Bipolar Disorder
* Type I diabetes mellitus or Type II diabetes mellitus requiring pharmacotherapy
* History of alcohol or drug abuse, current or within 5 years
* History of bulimia or anorexia nervosa
* History of surgical intervention for obesity
* History of seizure disorder or predisposition to seizures (e.g., history of cerebrovascular accident, significant head trauma, brain surgery, skull fracture, subdural hematoma, or alcohol withdrawal or febrile seizures)
* History of hypersensitivity to sulfonamides ("sulfa"), bupropion, or zonisamide
* History of nephrolithiasis (renal calculi)
* History of treatment with bupropion SR (Wellbutrin, Zyban) or zonisamide (Zonegran) within 12 months
* Use of drugs, herbs, or dietary supplements known to significantly affect body weight or participation in a weight loss management program within one month prior to baseline
* Loss or gain of more than 4.0 kilos within 3 months
* Women of child bearing potential not adhering to an acceptable form of contraception
* Pregnant or breast-feeding women
* Use of investigational drug, device or procedure within 30 days
* Participation in any previous clinical trial conducted by Orexigen Therapeutics
* Planned surgical procedure that can impact the conduct of the study
* Any condition which in the opinion of the investigator makes the subject unsuitable for inclusion in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 611 (Actual)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
% change in total body weight as measured between baseline and week 24 (ITT-LOCF analysis) | Baseline to week 24

SECONDARY OUTCOMES:
Absolute change in total body weight in kg. | Baseline to week 24
Proportion of subjects achieving > 5% weight loss. | Baseline to week 24
Proportion of subjects achieving > 10% weight loss. | Baseline to week 24
Proportion of subjects achieving > 5% weight loss at week 24 who maintain response to week 48 | Baseline to week 24
Change in measures of quality of life, sleep quality and sleep quantity | Baseline to week 24
Change in fasting triglycerides level | Baseline to week 24
Change in fasting blood glucose | Baseline to week 24
Change in systolic and diastolic blood pressure | Baseline to week 24
Change in HAMD-17 Maier subscale scores | Baseline to week 24
Change in Brief Assessment of Cognition composite scores | Baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Frank Greenway, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (15):
- United States (15):
  - SelfCenter, PC, Fairhope, Alabama
  - UCLA Center for Human Nutrition, Los Angeles, California
  - Scripps Clinic Del Mar, San Diego, California
  - Center for Human Nutrition University of Colorado Health Sciences Center, Denver, Colorado
  - George Washington University Weight Management Program, Washington D.C., District of Columbia
  - CSRA Partners in Health, Inc, Augusta, Georgia
  - Springfield Diabetes and Endocrine Center, Springfield, Illinois
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Nutrition and Weight Mangement Center Boston Medical Center, Boston, Massachusetts
  - Center for Nutrition and Metabolic Diseases, Reno, Nevada
  - Comprehensive Weight Control Program, New York, New York
  - Center for Nutrition and Preventive Medicine, Charlotte, North Carolina
  - MUSC Weight Mnagement Center, Charleston, South Carolina
  - The Cooper Institute, Dallas, Texas
  - Baylor Endocrine Center, Dallas, Texas